CLINICAL TRIAL: NCT01176058
Title: A Phase Iiib, Open-label, Randomized, Multi-center Study Of The Efficacy And Safety Of Anidulafungin Vs. Fluconazole, In The Treatment Of Subjects With Candidemia And/or Other Forms Of Invasive Candidiasis
Brief Title: A Study Of The Efficacy And Safety Of Anidulafungin Vs. Fluconazole In The Treatment Of Patients With Candidemia And/Or Other Forms Of Invasive Candidiasis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: A8851023
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-08

CONDITIONS: Candidemia
Keywords: Phase 3b; Efficacy and Safety evaluation of Anidulafungin; ICC
MeSH Terms: conditions — Candidemia | interventions — Anidulafungin; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Active Comparator)
  Interventions: Drug: Anidulafungin/Fluconazole

INTERVENTIONS:
Drug: Anidulafungin/Fluconazole — Anidulafungin:IV,100 mg daily preceded by an initial 200 mg dose on Day 1, 14 - 42 days Fluconazole: IV/Oral, 400mg,QD,14 - 42 days

SUMMARY:
In the treatment of patients with candidemia and/or other forms of invasive candidiasis , Anidulafungin is at least as effective and safe as Fluconazole.

DETAILED DESCRIPTION:
To support anidulafungin NDA in China Due to the challenges in subject recruitment resulting in protracted study course, Pfizer Inc. has decided to terminate trial A8851023 prematurely based on the recommendation by the senior management team on November 8, 2011. The decision to terminate the trial was not based on any safety concerns. All investigators were verbally informed by the study team since November 8, 2011 to stop the subject recruitment as soon as possible. All 17 enrolled subjects have been followed up on safety issues and no safety concerns were present by the data of these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Presence of candidemia or invasive candidiasis.
* Presence of one or more of signs and symptoms of acute fungal infection.

Exclusion Criteria:

* Subjects who received greater than 48 hours of systemic antifungal treatment for the Candida infection for which they will be enrolled.
* Subjects with hypersensitivity to echinocandins or azole therapy or drug excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- China (7):
  - Nanfang Hospital, Guangzhou, Guangdong
  - Nanjing General Hospital of Nanjing Military Command/Respiratory Department, Nanjing, Jiangsu
  - Changhai Hospital, Hemotology Department, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Medical School of Zhejiang University/Department of Hematology, Hangzhou, Zhejiang
  - Sir run run shaw hospital, Affiliated with school of medicine, Zhejiang University, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital / Department of Infectious Disease, Beijing
  - Institute of Antibiotics, Hua Shan Hospital, Fudan University, Shanghai

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851023&StudyName=A%20%20Study%20Of%20The%20Efficacy%20And%20Safety%20Of%20Anidulafungin%20Vs.%20Fluconazole%20In%20The%20Treatment%20Of%20Patients%20With%20Candidemia%20And/Or%20Other%20Forms

RESULTS

PARTICIPANT FLOW:
Groups:
- Anidulafungin: Intravenous (IV) Anidulafungin loading dose of 200 mg on Day 1 and then 100 mg daily from Day 2. Participants who completed a minimum of 7 days of IV treatment may have continued with IV treatment or may have been switched to oral fluconazole 400 mg daily up to a maximum of Day 42.
- Fluconazole: IV fluconazole 400 mg daily dose from Day 1 (dose reduction according to the participant's tolerability). Participants who completed a minimum of 7 days of IV treatment may have continued with IV treatment or may have been switched to oral fluconazole 400 mg daily up to a maximum of Day 42.
Period: Overall Study
Arm/Group | Anidulafungin | Fluconazole
Started | 9 | 8
Completed | 5 | 5
Not Completed | 4 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Insufficient clinical response | 2 | 2
Not completed — Insufficient mycological response | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anidulafungin | Fluconazole | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 1 | 4 | 5
  Between 45 and 64 years | 4 | 2 | 6
  More than 65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 8 | 5 | 13
Presence of Signs and Symptoms of Candidemia [Number; unit: participants] — Each participant could have been counted in more than 1 category for the signs and symptoms of Candidemia.
  participants
    Fever | 7 | 7 | 14
    Hypothermia | 0 | 0 | 0
    Tachycardia | 3 | 2 | 5
    White blood cell count decreased | 2 | 0 | 2
    White blood cell count increased | 3 | 1 | 4
    White blood cell morphology abnormal | 0 | 1 | 1
    Respiratory rate increased | 2 | 1 | 3
    Partial pressure of carbon dioxide (PCO2) decrease | 0 | 1 | 1
    Mechanical ventilation | 1 | 1 | 2
    Swelling | 1 | 2 | 3
    Feeling hot | 4 | 4 | 8
    Localized erythema | 1 | 0 | 1
    Purulence | 1 | 2 | 3
    Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Global Response at End of Intravenous Treatment (EOIT)
Description: Global response included clinical and microbiological success or failure. Success - clinical success (defined as the resolution or significant improvement in signs and symptoms of invasive candidiasis) and microbiological success (defined as the eradication of Candida species present at baseline, as determined on follow-up culture, or the presumed eradication, if culture data were not available [N/A] for a participant with a successful clinical response).
  Failure - Any case that did not meet the criteria for success.
Time Frame: End of Intravenous Treatment (Up to Day 42)
Population: Modified Intent-to-Treat (MITT) population: participants had confirmed diagnosis of candidemia or other forms of invasive candidiasis, received at least 1 dose of study medication treatment, had at least 1 post-baseline efficacy evaluation. N=number of participants with evaluable data; participants with missing or indeterminate data set to Failure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 8 | 7
percentage of participants
  Success | 62.50 [29.0 to 96.0] | 71.43 [38.0 to 100.0]
  Failure | 37.50 [4.0 to 71.0] | 28.57 [0.0 to 62.0]

2. Secondary Outcome: Percentage of Participants With Global Response at End of Treatment (EOT)
Description: Global response included clinical and microbiological success or failure. Success - clinical success (defined as the resolution or significant improvement in signs and symptoms of invasive candidiasis) and microbiological success (defined as the eradication of Candida species present at baseline, as determined on follow-up culture, or the presumed eradication, if culture data were N/A for a participant with a successful clinical response).
  Failure - Any case that did not meet the criteria for success.
Time Frame: End of Treatment (Up to Day 42)
Population: MITT population. N=number of participants with evaluable data; participants with missing or indeterminate data set to Failure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 8 | 7
percentage of participants
  Success | 62.50 [29.0 to 96.0] | 42.86 [6.2 to 79.5]
  Failure | 37.50 [4.0 to 71.0] | 57.14 [20.5 to 93.8]

3. Secondary Outcome: Percentage of Participants With Clinical Response at EOIT
Description: Clinical response included success and failure. Success included Cure (resolution of signs and symptoms of the Candida infection) and Improvement (significant, but incomplete resolution of signs and symptoms of Candida infection). Failure defined as No significant improvement in signs and symptoms or death due to Candida infection or circumstances prevented an evaluation from being made.
Time Frame: End of Intravenous Treatment (Up to Day 42)
Population: MITT population. N=number of participants with evaluable data; participants with missing data set to Failure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 8 | 7
percentage of participants
  Success | 75.00 [45.0 to 100.0] | 71.43 [38.0 to 100.0]
  Failure | 25.00 [0.0 to 55.0] | 28.57 [0.0 to 62.0]

4. Secondary Outcome: Percentage of Participants With Clinical Response at EOT
Description: as for outcome 3
Time Frame: End of Treatment (Up to Day 42)
Population: MITT population. N=number of participants with evaluable data; participants with missing data set to Failure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 8 | 7
percentage of participants
  Success | 75.00 [45.0 to 100.0] | 57.14 [20.5 to 93.8]
  Failure | 25.00 [0.0 to 55.0] | 42.86 [6.2 to 79.5]

5. Secondary Outcome: Percentage of Participants With Clinical Response at Follow-Up
Description: as for outcome 3
Time Frame: Post treatment follow-up visit (Up to Day 52)
Population: MITT population. N=number of participants with evaluable data; participants with missing data set to Failure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 8 | 7
percentage of participants
  Success | 75.00 [45.0 to 100.0] | 57.14 [20.5 to 93.8]
  Failure | 25.00 [0.0 to 55.0] | 42.86 [6.2 to 79.5]

6. Secondary Outcome: Percentage of Participants With Microbiological Response at EOIT
Description: Microbiological Success implies Eradication: culture negative for all Candida species present at baseline (documented), or culture data N/A (presumed). Microbiological Failure implies (1) Persistence: baseline Candida species present in repeat cultures (documented), or culture data N/A (presumed); (2) Recurrence: baseline Candida species isolated following eradication (documented), or culture data N/A (presumed); or (3) Indeterminate: culture data N/A (loss to follow-up or death that was not due to candidiasis or candidemia).
Time Frame: End of Intravenous Treatment (Up to Day 42)
Population: MITT population. N=number of participants with evaluable data; participants with missing or indeterminate data are set Failure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 8 | 7
percentage of participants
  Success | 75.00 [45.0 to 100.0] | 85.71 [59.8 to 100.0]
  Failure | 25.00 [0.0 to 55.0] | 14.29 [0.0 to 40.2]

7. Secondary Outcome: Percentage of Participants With Microbiological Response at EOT
Description: as for outcome 6
Time Frame: End of Treatment (Up to Day 42)
Population: MITT population. N=number of participants with evaluable data; participants with missing or indeterminate data are set to Failure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 8 | 7
percentage of participants
  Success | 75.00 [45.0 to 100.0] | 57.14 [20.5 to 93.8]
  Failure | 25.00 [0.0 to 55.0] | 42.86 [6.2 to 79.5]

8. Secondary Outcome: Percentage of Participants With Microbiological Response at Follow-Up
Description: as for outcome 6
Time Frame: Post treatment follow-up visit (Up to Day 52)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 8 | 7
percentage of participants
  Success | 62.50 [29.0 to 96.0] | 57.14 [20.5 to 93.8]
  Failure | 37.50 [4.0 to 71.0] | 42.86 [6.2 to 79.5]

9. Secondary Outcome: Number of Participants Who Died
Time Frame: Baseline to Day 52
Population: Safety population: All participants who have received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 9 | 8
participants | 1 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Anidulafungin | Fluconazole
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/8
Other Adverse Events (participants affected / at risk) | 6/9 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=9) | Fluconazole (N=8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=9) | Fluconazole (N=8)
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Intestinal obsturction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Chest discomfort (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to small enrollment, the per-protocol population was not determined, and analysis was performed on the mITT population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.